CLINICAL TRIAL: NCT03705897
Title: PROSPR Project 1: Identifying and Tracking Personalized CRC Screening Regimens for Patients in Clinical Settings
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Celette Skinner, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 102011-068; STU 102011-068 (Other: UT Southwestern Medical Center)
Record Dates: First submitted 2017-02-09; First posted 2018-10-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: ColoRectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening (Other): Employ innovative methods for assessing personalized guideline-based screening in the clinic setting to evaluate guideline-based, over- and under-screening. Interventions include Computerized Risk Stratification Tool, Algorithmic Risk Stratification Tool, and Step completion assessment.
  Interventions: Other: Computerized Risk Stratification Tool; Other: Algorithmic Risk Stratification Tool; Other: Step completion assessment

INTERVENTIONS:
Other: Computerized Risk Stratification Tool — Implement a novel computerized risk stratification tool in Parkland community-oriented primary-care clinics that collects data directly from patients and uses a computerized algorithm system to generate their personalized guideline-based next steps in the screening regimen
Other: Algorithmic Risk Stratification Tool — Implement a novel algorithmic risk stratification system in Parkland's endoscopy clinics that, based on test findings entered by colonoscopists, generates personalized guideline-based next steps in the screening regimen for patients with colorectal polyps removed at olonoscopy
Other: Step completion assessment — Assess completion of guideline-recommended steps in personalized screening regimens, under-screening, and over-screening

SUMMARY:
The overall goal of the Parkland-UT Southwestern Population-based Research Optimizing Screening through Personalized Regimens (PROSPR) Center is to optimize colon cancer screening through personalized regimens in the integrated safety-net clinical provider network, which serves a large and diverse population of under- and un-insured patients in Dallas. Together, three research projects will assess clinic, system, and organizational factors associated with over-, under- and guideline-based screening among this important population and will compare benefits, harms, and costs of strategies for facilitating optimized screening regimens. The theme of optimizing colorectal cancer screening in a safety-net clinical provider network brings together several components. Its focus on colorectal cancer (CRC) screening which is important, because CRC is the second cancer killer in the US while being the only major cancer for which optimized screening results in primary prevention. Despite this strong potential benefit, CRC screening remains suboptimal overall, and especially among low-income and minority individuals served by safety-nets. Safety-net networks therefore offer tremendous potential for CRC prevention and control, but numerous factors at the clinics-, system-, and organization-level influence their ability to provide optimized care.

DETAILED DESCRIPTION:
Each of the Population-based Research Optimizing Screening through Personalized Regimens (PROSPR) Center's projects is innovative and addresses the continuum of care. Project 1 addresses transitions 1 and 3, employing novel, algorithmically driven tools in clinics to determine personalized optimized screening regimens for individual patients and track whether each has received the indicated guideline-based screening. Project 2 addresses all three transitions through a novel comparative effectiveness study of benefits, risks, and costs of two outreach strategies for promoting screening completion and guideline-appropriate follow-up. Project 3 addresses transitions 2 and 3 by focusing on organizational culture, structure, and protocols, using both quantitative and qualitative methods to elucidate factors influencing completion of effective screening processes. These projects address research priorities identified through a recent National Institute of Health (NIH) State of the Science Conference, including: implementing interventions proven effective at increasing colorectal cancer (CRC) screening (Projects 1 & 2), conducting research to assess effectiveness of tailoring programs to match characteristics and preferences of target populations (Project 1), implementing systems to ensure follow up of positive CRC screening results (Projects 1, 2 & 3), and conducting studies to determine comparative effectiveness of CRC screening methods in usual practice (Project 2).

PROSPR Center's goals are to:

1. Develop a Parkland-UT Southwestern PROSPR Center to promote coordinated, transdisciplinary research to evaluate and improve the CRC screening process in a large population-based safety-net.
2. Conduct three projects that address the continuum of care for CRC screening and address these goals:

   Project 1- Employ innovative methods for assessing personalized guideline-based screening in the clinic setting to evaluate guideline-based, over- and under-screening; Project 2 - Compare benefits, harm, and costs of three system-level strategies for inviting patients to screening and promoting guideline-based follow up, with particular focus on completing an effective screening process.

   Project 3 - Examine specific organizational factors that contribute to completion of guideline-based screening processes and examine which organizational factors modify relationships between social disadvantage and completion of guideline-based repeat screening and follow up of abnormal test results.
3. Contribute to a national PROSPR network by actively participating in network activities, including:

   1. collaborating with the National Data Coordinating Center regarding approaches for measuring screening effectiveness, (b) sharing algorithmically driven tools facilitating personalized screening regimes, (c) sharing electronic medical record (EMR) capabilities with other Epic institutions, and (d) becoming a leader in cancer screening processes in safety-net systems. While the SPDU will be exclusively responsible for all required PROSPR network data collection, processing and transfer activities, our complementary Shared Research Resources Core (SRRC) will serve as the local "data coordinating center" of our PROSPR center. The SRRC will work with Projects 1-3 to identify patients for recruitment; track study accrual; and manage, process, and analyze all Project data. The SRRC will also help assure consistent data definitions and terminology for harms, benefits, and other common domains across the screening process documentation unit (SPDU) and Projects. The SRRC and SPDU will work closely together as much of the required SPDU screening process data will be used by the SRRC to identify eligible patients for Projects 1-3, and ascertain the processes and outcomes of the CRC screening process for study participants. An innovative activity of the SRRC will be to extract from Epic a novel set of electronically derived measures of social disadvantage previously developed by the Parkland Center for Innovation.27 This will empower Projects 1 and 2 to examine the influence of these factors on the in-reach and out-reach programs, as well as provide Project 3 with critical explanatory variables to understand the impact of clinic-level organizational factors on the CRC screening process.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ages 25-64, presenting for appointment will be eligible to participate.
* Patients 25-49 must also have family hx of CRC or personal hx of inflammatory bowel disease or adenomatous polyps.
* No racial or ethnic group will be excluded from participation.
* Both English and Spanish speakers will be eligible for participation.

Exclusion Criteria:

* Patients with a personal history of CRC are not eligible to participate.
* Patients who do not speak Spanish or English or have severely impaired hearing or speech or do not give informed consent will also be excluded from participation.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9865 (Estimated)
Dates: Start 2013-08; Primary Completion 2025-12-27 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving appropriate screening regimen. | Three years
  Proportion of patients achieving appropriate screening regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Celette Skinner, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No